CLINICAL TRIAL: NCT00537108
Title: BRIDGES: A Randomized Trial of Community-Based Care Management For Teen/Young Adult Mothers and Fathers
Brief Title: Community-Based Care Management For Teen/Young Adult Mothers and Fathers
Acronym: BRIDGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: UMB School of Medicine Department of Family and Community Medicine (Unknown); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beth Barnet, Professor, Family and Community Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H-29138
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Pregnancy
Keywords: Pregnancy in adolescence
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Intervention Model Description: Motivational intervention and support
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HV (Experimental): Intervention arm.
  Interventions: Behavioral: Home visiting and care management
- Cntr (No Intervention): Usual care control

INTERVENTIONS:
Behavioral: Home visiting and care management — Third trimester teens are assigned a Care Manager (CM) who establishes a continuity relationship and provides monthly visits until the index child is 2 years old. Core services for intervention group include: 1)Baseline and ongoing assessment of health, mental health, housing, daycare, and school needs; 2)Administration of a culturally sensitive, developmentally relevant parenting curriculum; 3)Computer Assisted Motivational Interviewing to promote healthy relationships, improve contraceptive practices, focus on goals, and promote school continuation; 4)Efforts to engage the young father; 5)Linkage and coordination with primary care for teen, child, young father; 6)Support & skills-building for school continuation, higher education, and job readiness.
  Arms: HV

SUMMARY:
Teenagers who become parents often struggle with new challenges as they try to take care of their children and themselves. Programs that provide teens with support, education, and counseling may help teens to become the best parents they can be and reach their own goals. Health care providers who take care of pregnant and parenting teenagers are trying to find out what types of programs are most helpful for the physical, emotional, and social health of pregnant and parenting teenagers. The purpose of this study is to find out what kinds of activities help teens be successful as parents and achieve success in their lives.

DETAILED DESCRIPTION:
Pregnant teenagers and teenagers who have children less than 2 weeks old and who attend either University Family Medicine, the Maryland Women's Center, Teen Tot Clinic, University Care at Edmonson Village, Weinberg Community Health Center, or Maryland General Outpatient clinics will be asked to participate in a home visiting and care management program and study. Those agreeing to participate are placed into one of two groups. One group receives a Home Visiting and Care Management Program along with their usual medical care. The other group receives only their usual medical care.

If placed into the home visiting group, the teen is given a home visitor (also called a Care Manager). The Care Manager arranges to meet with the teen every month until the teen's baby is 2 years old. The meetings last about 1 hour and usually take place in the teen's home.

The Care Manager provides 4 Core Services to the teen:

1. Baseline and ongoing monthly needs assessment for healthcare, mental health, school/job attainment, daycare, housing stability;
2. Computer Assisted Motivational Interviewing (CAMI) sessions with teen mother. In CAMI sessions, the teen answers questions on a laptop computer that assess partner relationships, sexual behaviors, & risk for repeat pregnancy. Following the assessment, the trained Care Manager conducts motivational interviewing, a counseling technique aimed at assisting the teen to improve contraceptive and condom use, focus on goals, and promote school continuation;
3. Parenting instruction with a culturally sensitive, developmentally relevant parenting curriculum; and
4. Coordination and linkage with primary care and community partners (e.g. UMB Division of Community Psychiatry) with respect to health care, mental health care, and other services.

If the teen grants permission, we will try to contact her baby's father and invite him to participate in similar activities.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant teenagers
* Ages 12-18 years old
* >= 24 weeks gestation
* Attending any of 5 West Baltimore prenatal care sites.
* Male partner (baby's father) if the pregnant teenager agrees to let the program contact him to invite participation.

Exclusion Criteria:

* Age < 18 years and no parent/guardian able to grant consent.
* Male partner of a pregnant teen/teen mother if she does not grant consent to let us contact him and invite participation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Repeat pregnancy | Within 2 years of the index birth
Parenting attitudes and behaviors | at 1 year and 2 years postpartum
School continuation or graduation | at 2 years postpartum

SECONDARY OUTCOMES:
Remission of depression | at 1 year and 2 years postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Beth Barnet, M.D., Principal Investigator — University of Maryland
Locations (1):
- UMB School of Medicine Department of Family and Community Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No